CLINICAL TRIAL: NCT06874400
Title: Comparison of Dairy and Plant-based Alternatives in Adolescents and Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 47896; 72072239 (Other Grant/Funding Number: Dairy Farmers of Canada)
Record Dates: First submitted 2025-03-04; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Glycemic Response to Feeding in Healthy Participants; Postprandial Amino Acid Concentrations; Appetite Regulation
Keywords: Nutrition; dairy; plant-based foods; glycemic response; appetite; protein; food; adolescents; older adults; overweight
MeSH Terms: conditions — Overweight | interventions — Milk; Yogurt; Cheese; Whey; Meat Substitutes; Soy Milk; Soy Foods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dairy (Experimental): Participants will consume 2 servings of a commerically available dairy product.
  Interventions: Other: Dairy
- Plant-based alternative (Experimental): Participants will consume 2 servings of a commercially available plant-based alternative product.
  Interventions: Other: Plant-based alternative

INTERVENTIONS:
Other: Dairy — The dairy products that participants will be required to consume include: 1) Trial 1: 2% cow's milk; 2) Trial 2: dairy yogurt; 3) Trial 3: 2% cottage cheese; 4) Trial 4: 2% cow's milk; and 5) Trial 5: isolated whey protein beverage. Participants will only be enrolled in 1 of the 5 trials; as such, they will only consume the 1 dairy product in that trial.
  Other Names: Milk; yogurt; cheese; whey
  Arms: Dairy
Other: Plant-based alternative — The plant-based products that participants will be required to consume include: 1) Trial 1: soy beverage; 2) Trial 2: plant-based yogurt; 3) Trial 3: tofu; 4) Trial 4: 2% simulated milk; and 5) Trial 5: isolated soy protein beverage. Participants will only be enrolled in 1 of the 5 trials; as such, they will only consume the 1 plant-based alternative product in that trial.
  Other Names: soy beverage; plant-based yogurt; simulated milk; soy; tofu
  Arms: Plant-based alternative

SUMMARY:
The purpose of the Dairy vs Plant study is to compare the effects of dairy and plant-based alternative products on blood sugar regulation and nutrient quality in adolescents and older adults. We are inviting healthy, non-diabetic participants aged 14-18 and 60-75, both males and females to participate. The study will take place in the Nutrition Intervention Center located at the Department of Nutritional Sciences, University of Toronto St. George campus. Participants will be asked to come to the Nutrition Intervention Center on 3 separate occasions: once for an in-person screening lasting approximately 30min and 2 times for study visits lasting approximately 2.5 hrs each. The entire study will take a minimum of 2 weeks to complete. You will be asked to fast for 12hrs (overnight) prior to each study visit. You will also be instructed to maintain the same dietary and sleep patterns, refrain from exercise and alcohol consumption the days before the study visits. During these study visits, you will be asked to consume either a dairy or a plant-based alternative product, as well as a pizza meal. You will periodically fill out questionnaires rating your feelings and perceptions and provide blood samples through finger pricks and intravenously through forearm to measure blood sugar, insulin, hormones, and amino acids. You will be compensated for your time and travel expenses.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-18 years old (adolescents) or 60-75 years old (older adults)
* BMI z-score >+1SD, <+2SD (adolescents) or BMI 25-30 kg/m2 (older adults)
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the study.
* Willing to maintain current dietary supplement use throughout the study. On study visit days, subject agrees not to take any supplements until dismissal from the Nutrition Intervention Center.
* Willing to abstain from alcohol consumption for 24hrs prior to all study visits.
* Willing to avoid vigorous physical activity for 24hrs prior to all study visits.
* Willing to refrain from cannabis use throughout the entire duration of the study.
* Willing to refrain from protein supplement use (e.g. protein powder) throughout the entire duration of the study.
* Understands the study procedures, provides informed consent to participate in the study, and authorizes release of relevant protected health information to the study investigator.

Exclusion Criteria:

* Smoking
* Thyroid problems
* Lactose intolerance and/or allergies, intolerances, or sensitivities to study treatments
* Previous history of cardiovascular disease, diabetes, liver or kidney disease, inflammatory bowel disease, celiac disease, short bowel syndrome, malabsorptive syndrome, pancreatitis, gallbladder or biliary disease
* Presence of gastrointestinal disorder or surgeries within the past year.
* Inability to comply with the experimental procedures and follow our safety guidelines
* Regular breakfast skipping (>3 days a week)
* On a special diet (e.g. ketogenic, Atkins, high protein) or restrained eaters as identified by a score of >20 on the Eating Attitudes Questionnaire
* Difficulties with eating or swallowing
* Fasting blood glucose >5.6mmol/L measured at screening
* Uncontrolled hypertension (systolic blood pressure >120mmHg, diastolic blood pressure >80mmHg) as defined by the average blood pressure measured at screening
* Weight gain or loss of >10lbs in previous three months
* Consuming prescription or non-prescription drug, herbal or nutritional supplements known to affect outcome of the study as per investigator's judgement

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | Over 145 minutes after treatment consumption at each session, for a total of 2 weekly sessions.
  Blood glucose will be measured via finger-prick using a glucose meter at 0, 20, 35, 50, 65, 95, 125, and 145 minutes after treatment consumption.

SECONDARY OUTCOMES:
Insulin | Over 145 minutes after treatment consumption at each session, for a total of 2 weekly sessions.
  Insulin will be measured in the plasma through intravenous blood collection at 0, 35, 65, 95, 125, and 145 minutes after treatment consumption.
Glucagon-like Peptide-1 (GLP-1) | Over 145 minutes after treatment consumption at each session, for a total of 2 weekly sessions.
  GLP-1 will be measured in the plasma through intravenous blood collection at 0, 35, 65, 95, 125, and 145 minutes after treatment consumption.
Glucagon-like Peptide-2 (GLP-2) | Over 145 minutes after treatment consumption at each session, for a total of 2 weekly sessions.
  GLP-2 will be measured in the plasma through intravenous blood collection at 0, 35, 65, 95, 125, and 145 minutes after treatment consumption.
Gastric Inhibitory Polypeptide (GIP) | Over 145 minutes after treatment consumption at each session, for a total of 2 weekly sessions.
  GIP will be measured in the plasma through intravenous blood collection at 0, 35, 65, 95, 125, and 145 minutes after treatment consumption.
Leptin | Over 145 minutes after treatment consumption at each session, for a total of 2 weekly sessions.
  Leptin will be measured in the plasma through intravenous blood collection at 0, 35, 65, 95, 125, and 145 minutes after treatment consumption.
Peptide YY (PYY) | Over 145 minutes after treatment consumption at each session, for a total of 2 weekly sessions.
  PYY will be measured in the plasma through intravenous blood collection at 0, 35, 65, 95, 125, and 145 minutes after treatment consumption.
Cholecystokinin (CCK) | Over 145 minutes after treatment consumption at each session, for a total of 2 weekly sessions.
  CCK will be measured in the plasma through intravenous blood collection at 0, 35, 65, 95, 125, and 145 minutes after treatment consumption.
Ghrelin | Over 145 minutes after treatment consumption at each session, for a total of 2 weekly sessions.
  Ghrelin will be measured in the plasma through intravenous blood collection at 0, 35, 65, 95, 125, and 145 minutes after treatment consumption.
Adiponectin | Over 145 minutes after treatment consumption at each session, for a total of 2 weekly sessions.
  Adiponectin will be measured in the plasma through intravenous blood collection at 0, 35, 65, 95, 125, and 145 minutes after treatment consumption.
Amino Acids | Over 145 minutes after treatment consumption at each session, for a total of 2 weekly sessions.
  Amino acid concentrations will be measured in the plasma through intravenous blood collection at 0, 35, 65, 95, 125, and 145 minutes after treatment consumption.

OTHER OUTCOMES:
Appetite | Over 145 minutes after treatment consumption at each session, for a total of 2 weekly sessions.
  Appetite will be assessed through Adaptive Visual Analogue Scales (AVAS) questionnaires completed at 0, 20, 35, 50, 65, 95, 125 and 145 minutes after treatment consumption, and through an ad libitum pizza meal provided at 125 minutes post-treatment consumption, where participants will be instructed to eat until they are comfortably full over 20 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: G. Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- Nutrition Intervention Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared, as all data will be de-identified and pooled during the analysis. Only researchers directly involved in the study will have access to the data.

REFERENCES:
- [Background] Da Silva N, Anderson G, Amr A, Vien S, Fabek H. A comparison of the effects of dairy products with their plant-based alternatives on metabolic responses in healthy young Canadian adults: a randomized crossover study. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-17. doi: 10.1139/apnm-2024-0158. PMID 39146559